CLINICAL TRIAL: NCT06839690
Title: Comparison of Sub-maximal Voluntary Isometric Training vs Eccentric Training in Management of De Quervain Tenosynovitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/1
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: De Quervain Syndrome
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sub-maximal Voluntary Isometric training Group (Active Comparator): Group A will recieve ultrasound therapy for symptoms management and isometric training of thumb muscles (abducttor pollices longus and extensor pollices brevis) to gain improvement in range of motion and strength
  Interventions: Procedure: Isometric training of thumb muscles; Procedure: Ultrasound
- Eccentric training Group (Experimental): Group B will receive the ultrasound therapy similar to group A for symptoms management and eccentric training of thumb muscles to gain improvement in range of motion and strength of thumb
  Interventions: Procedure: Eccentric training for thumb muscles; Procedure: Ultrasound

INTERVENTIONS:
Procedure: Isometric training of thumb muscles — Isometric training for thumb extension, abduction, radial and ulnar deviation will be performed in 3 sessions/ week for 4 weeks. The exercise protocol will begin with training using manual resistance and progress with training against resistance of elastic band and theraband.I
  Arms: Sub-maximal Voluntary Isometric training Group
Procedure: Eccentric training for thumb muscles — In Group B, eccentric training for thumb extension, abduction, radial and ulnar deviation will be performed in 3 sessions/ week for 4 weeks. The exercise protocol will begin with training using unweighted and weighted hammer curls and progress with training using elastic band, dumbbell and theraband.
  Arms: Eccentric training Group
Procedure: Ultrasound — Therapeutic ultrasound for symptom management

SUMMARY:
This study is a randomised control trial and the purpose of this study is to compare the effects of Sub-maximal Voluntary Isometric Training vs Eccentric Training in Management of De Quervain Tenosynovitis

DETAILED DESCRIPTION:
Participants will be recruited into their respective groups using a coin toss method. De Quervain Tenosynovitis will be assessed using the following tests:

1. Wrist hyperflexion and abduction of thumb (WHAT) test
2. Finkelstein's / Eichhoff's test
3. De Quervain Screening Tool

ELIGIBILITY:
Inclusion Criteria:

* Patients having history of pain, tenderness in thumb region from 3 weeks or more
* Age 21-50
* Both genders
* Individuals meeting the diagnostic criteria i.e.
* A score of 3 or more out of 7 on De Quervain screening tool.
* Positive Wrist hyperflexion and abduction of thumb (WHAT) test
* Positive Finkelstein's / Eichhoff's test

Exclusion criteria:

* Diagnosed cases of Osteoarthritis of 1st CMC joint and Rheumatoid arthritis
* C6 cervical radiculopathy
* Any systemic inflammatory condition like septic arthritis
* Carpal Tunnel Syndrome
* Complex regional pain syndrome
* Previous surgery impacting the first extensor compartment of the wrist
* Corticosteroid injection in the radial wrist region within 3 months of enrolment into the study
* If patient had undergone isometric thumb exercises or any strengthening protocol lasting greater than 2 weeks for the management of their current episode of de Quervain's syndrome

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Grip Strength measurement | 4 weeks
  Power grip strength will be measured using hand held dynamometer and pinch grip strength will be measured using Modified sphygmomanometer

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physcial Therapy, Rawalpindi, Punjab Province, Pakistan